CLINICAL TRIAL: NCT00551746
Title: Anti-thrombotic Effects of Long Term Consumption of Purple Grape Juice in Healthy People
Brief Title: The Purple Grape Juice Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Deseret Foundation (Other); Welch's, Inc. (Industry); ThromboVision, Inc. (Industry)
Responsible Party: Benjamin D. Horne, Intermountain Healthcare
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 128-126
Record Dates: First submitted 2007-10-29; First posted 2007-10-31 (Estimated); Results first posted 2011-09-07 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Cardiovascular Disease
Keywords: purple grape juice; antioxidants; platelet aggregation; anti-thrombotic
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Grape Juice
  Interventions: Dietary Supplement: Purple Grape Juice
- 2 (Placebo Comparator): Grape Juice Placebo
  Interventions: Dietary Supplement: Purple Grape Juice

INTERVENTIONS:
Dietary Supplement: Purple Grape Juice — Grape Juice

SUMMARY:
Coronary heart disease (CHD) is the largest contributor to morbidity and mortality in the Western world and is associated with high-calorie diet, high body mass, and a variety of other factors. CHD can lead to myocardial infarction (MI) and other embolic events. In some areas such as France, though, a paradox of high-cholesterol diets but low CHD and MI incidence have been found. This paradox has been traced to the consumption of red wine. Further research suggests that components of the grapes used in red wine may be the source of the cardio-protective factors that have resulted in the French paradox. These components are also present in purple grape juice (PGJ). PGJ has been shown to have a variety of potential cardio-protective effects, including inhibition of platelet aggregation. Since PGJ does not contain alcohol it may provide an additional benefit by avoiding the physical and social implications of alcohol abuse. Since most of the research of PGJ has been in vitro, though, and the few studies in vivo have been in cross-over studies and over very short durations of 7 to 14 days, additional research is required to determine whether the long-term consumption of PGJ is of additional and sustained benefit, similar to long-term use of red wine in France. The proposed study is a 2 arm randomized, controlled (double-blind) study of PGJ and a calorically-matching placebo drink in 100 healthy individuals.

DETAILED DESCRIPTION:
The study treatment period will be 90 days (13 weeks, or 3 months) and the treatment dose will be 7 mL/kg/day. The treatment dose is a standard dose previously worked out in other research and was used in a variety of other clinical research (27, 32). Study randomization will be performed in a double-blind fashion with study investigators and participants unaware of group assignment. Randomization order will be created using a randomized blocked design. After volunteer consent is provided, the clinical study coordinator will open a sequentially-numbered envelope containing the study group assignment and provide a 4 week supply of study beverage.

Participants will be seen for follow-up study visits at approximately 4 week intervals after the baseline enrollment visit. Compliance with study treatment (PGJ or placebo) will be assessed by interview at visits 2, 3, and 4. At the conclusion of visits 2 and 3, a supply of study beverage will be provided to the participant for consumption during the ensuing 4 weeks. Study beverage supplies remaining at the end of the 90-day study period will be donated to each participant.

Platelet Aggregation testing will be performed by ThromboVision (Salt Lake City, UT) using multiple platelet agonists, including ADP, collagen/epinephrine, PMA, and TRAP. Each of these aggregation inducers target a separate platelet activation pathway.

ELIGIBILITY:
Inclusion Criteria:

1. The volunteer (male or non-pregnant female, any ethnicity) must be > 18 years of age.
2. The volunteer has no history of a physician diagnosis of atherosclerosis such as carotid, peripheral, or coronary artery disease (CAD).
3. The volunteer has no history of a physician diagnosis of pulmonary embolism (PE), MI, or stroke.
4. The volunteer must sign a written informed consent, prior to the procedure, using a form that is approved by the local Institutional Review Board.

Exclusion Criteria:

1. A diagnosis if diabetes mellitus.
2. The limitations for specific medications, supplements and food items are exceeded as follows:

More than 1 normal dose of the following medications and/or supplements once a week during the 3 months prior to enrollment:

* aspirin • ibuprofen • fish-oil extracts
* antioxidants • vitamins

More than 1 normal serving per week in the 3 months prior to enrollment:

* other grape juices • tea • wine
* beer • alcoholic drinks • grapes

More than 5 servings per day in any combination in the 7 days (1 weeks prior to enrollment:

* non-grape juices • garlic • broccoli
* apples • any type of berries • onions Volunteer is pregnant or lactating at the time of enrollment.

Secondary Exclusions:

1. Use of any of the above listed items during the 12 week course of study treatment will be documented and excess use 3 times or more will result in an administrative withdrawal of the volunteer from the study prior to the measurement of the next monthly platelet aggregation laboratory values (although those values will be measured for exploratory evaluation and the participant will remain under treatment until the end of the 12 week period).
2. Routine consumption of fruit juices, or of >5 servings per day of referenced fruits or vegetables, will result in administrative withdrawal of the participant from the study's primary aim.
3. Although it is unlikely the use of PGJ or look alike/ taste alike (placebo) beverage will harm the pregnant or lactating woman, the dietary restrictions placed on the participant for the duration of the study may conflict with dietary recommendations for pregnant or lactating women. Women of child bearing potential, therefore, will meet a secondary exclusion if they become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-07; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Horne, PhD, MPH, Principal Investigator — Intermountain Medical Center, Murray, UT
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: August, 2007 to June, 2009
Groups:
- Grape Juice: 100% Grape Juice
- Grape Juice Placebo: Taste, color, and calorically matched grape juice placebo
Period: Overall Study
Arm/Group | Grape Juice | Grape Juice Placebo
Started | 36 | 34
Completed | 25 | 26
Not Completed | 11 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Grape Juice | Grape Juice Placebo | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 34 | 68
  >=65 years | 2 | 0 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 40.8 (14.1) | 42.3 (11.4) | 41.6 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 23 | 17 | 40
Region of Enrollment [Number; unit: participants]
  United States | 36 | 34 | 70

OUTCOME MEASURES:

1. Primary Outcome: Compare Change in Platelet Aggregation as Measured by Adenosine Diphosphate (ADP) Between PGJ and Placebo
Description: Platelet aggregation was measured using the agonist ADP (10 microM) in a light transmission aggregometer and compared between PGJ and placebo via the intent-to-treat paradigm.
Time Frame: 90-days
Population: The number of participants evaluated were those who had both a baseline and visit 4 platelet aggregation and platelet-dependant inflammatory marker values
Measure: Mean (Standard Deviation); unit: percent
Groups:
- Purple Grape Juice: 100% grape juice
- Placebo: Taste, color, and colorically matched grape juice placebo
Arm/Group | Purple Grape Juice | Placebo
Number analyzed (Participants) | 23 | 25
percent | 1.59 (16.2) | -12.3 (17.8)

2. Secondary Outcome: Compare Platelet Inhibitory Pathways of ADP,TRAP, PMA, Arachadonic Acid Between PGJ and Placebo.
Description: The platelet inhibitory pathway in which PGJ functions by performing platelet aggregation tests using agonists for the 4 major platelet activation pathways: ADP,thrombin receptor-activator peptide (TRAP), phorbol 12-myristate 13-acetate (PMA), arachadonic acid(10 microM) in a light transmission aggregometer and compared between PGJ and placebo via the intent-to-treat paradigm.
Time Frame: 90-days
Reporting Status: Not Posted
Measure: unit: percent

3. Secondary Outcome: The Impact of Polymorphism in Haemostatic Genes on Variation in Platelet Function Among Participants Based on Long-term PGJ Consumption.
Time Frame: 90-days
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: participants

ADVERSE EVENTS:
Arm/Group | Grape Juice | Grape Juice Placebo
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/34
Other Adverse Events (participants affected / at risk) | 0/36 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No